CLINICAL TRIAL: NCT05846360
Title: The Technical and Operational Performance of the QuidelOrtho Savanna RVP4 Analyzer
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0318; SMPH/FAMILY MED/CLINIC WINGRA (Other: UW Madison)
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Respiratory Viral Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Nasal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ORCHARDS Study Specimens: Archived ORCHARDS study specimens

SUMMARY:
The purpose of this study is for the research team to become familiar with and evaluate the technical and operational performance of the QuidelOrtho Savanna RVP4 analyzer by testing 120 archived specimens that were previously tested at the Wisconsin State Laboratory of Hygiene (WSLH) by RT-PCR and multiplex respiratory pathogen panel within the last year.

DETAILED DESCRIPTION:
To test the technical and operational performance of the QuidelOrtho Savanna RVP4 analyzer, the investigator proposes to test samples archived from the ORegon CHild Absenteeism due to Respiratory Disease Study (ORCHARDS) study (HSC 2013-1357), a study that had the goal to "develop and implement a system for daily school-based monitoring of ILI (influenza-like illness) and CLI (COVID-like illness) student absenteeism in kindergarten (K) through grade 12 schools, and assess the system's usability for early detection of accelerated influenza, SARS-CoV-2 and other respiratory pathogen transmission in schools and surrounding communities".

The deidentified paired (WSLH vs. Savanna RVP4) results will be used by QuidelOrtho Corporation to evaluate the technical and operational performance of the analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Previously collected specimens from the ORCHARDS study.

Exclusion Criteria:

* Specimens not collected as part of the ORCHARDS study.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: School-aged children
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Number of Samples with Matching Results | up to 6 months
  There were a number of viruses detected in the ORCHARDS study [Ad, adenovirus; CoV, coronavirus; Flu, influenza virus; hMPV, human metapneumovirus; PIV, parainfluenza virus; R/E, rhinovirus/enterovirus; RSV, respiratory syncytial virus]. Reported here are the number of samples for which the Savanna RVP4 results match the WSLH results.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Temte, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Temte JL, Barlow S, Goss M, Temte E, Bell C, He C, Hamer C, Schemmel A, Maerz B, Comp L, Arnold M, Breunig K, Clifford S, Reisdorf E, Shult P, Wedig M, Haupt T, Conway J, Gangnon R, Fowlkes A, Uzicanin A. The Oregon Child Absenteeism Due to Respiratory Disease Study (ORCHARDS): Rationale, objectives, and design. Influenza Other Respir Viruses. 2022 Mar;16(2):340-350. doi: 10.1111/irv.12920. Epub 2021 Oct 8. PMID 34623760